CLINICAL TRIAL: NCT06780839
Title: Postoperative Adjuvant Treatment of ALK-positive Non-small Cell Lung Cancer with Ensartinib Guided by MRD: a Single-arm, Multicenter Study
Brief Title: Adjuvant Treatment of ALK-positive Non-small Cell Lung Cancer with Ensartinib Guided by MRD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Collaborators: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Wu Nan, Professor, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BD-EN-IV025
Record Dates: First submitted 2024-12-29; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-12

CONDITIONS: NSCLC, Stage I, II, IIIA, IIIB
Keywords: NSCLC; ALK positive; MRD; adjuvant therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — ensartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ensartinib (Experimental)
  Interventions: Drug: Ensartinib

INTERVENTIONS:
Drug: Ensartinib — Patients will receive Ensartinib 225mg QD by MRD test guided, if MRD test shows negative, only ensartinib will be given. if MRD test turns from negative to posive, patients will receive step-up treatment, which is ensartibe plus platinum - based doublet chemotherapy no more than 4 cycles. If MRD test turns from posive to negative, only ensartinib will be given. if MRD test constantly shows positive, MDT will determine the next step ensartib-based therapy.

SUMMARY:
To explore the efficacy and safety of ensartinib on adjuvant therapy guided by MRD in IA3-IIIB (T3N2) stage ALK-positive non-small cell lung cancer patients.

DETAILED DESCRIPTION:
Eligible subjects will take ensartinib 225 mg once daily. Postoperative tissues will be collected for customized minimal residual disease (MRD) detection (tumor-informed MRD). MRD tests will be conducted within 14 to 50 days after surgery (before adjuvant therapy), every 12 weeks ± 7 days for the first two years, and every 24 weeks ± 7 days for the third year. Subjects with negative MRD after surgery will receive ensartinib treatment. If MRD turns positive, they will receive ensartinib 225 mg QD combined with platinum-based doublet chemotherapy (2 to 4 cycles) as a step-up treatment. Subjects with positive MRD after surgery will also receive ensartinib treatment. If MRD remains positive at the next MRD test, they will receive ensartinib 225 mg QD combined with platinum-based doublet chemotherapy (2 to 4 cycles) as a step-up treatment. If MRD turns negative during treatment, ensartinib monotherapy will be resumed. If MRD turns positive again, the subsequent treatment mode will be determined by the MDT discussion group composed of the main center researchers, including but not limited to monotherapy or combination with platinum-free chemotherapy until 3 years, or MRD turns negative, or intolerable toxicity, or radiological recurrence, whichever occurs first. For patients who remain MRD positive after 3 years of treatment, the MDT group will discuss the next steps.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed primary non-small cell lung cancer;
2. Age ≥18 years old, gender unlimited;
3. The stage of the disease was based on AJCC/UICC 8th edition of lung cancer staging criteria; Complete surgical resection (R0) of primary lung cancer with Stage IA3 with high-risk recurrence factors, stage IB, II, IIIA, and IIIB (T3N2M0 only) of non-small cell lung were pathological confirmed;
4. Full recovery from surgery;
5. The biopsy or postoperative tumor tissue samples tested by the local laboratory are positive for ALK, and can be accepted by IHC, RT-PCR, FISH and NGS test results;
6. Intended to receive enshatinib postoperative adjuvant therapy;
7. ECOG physical status score is 0-1;
8. Has good hematopoietic and organ function, and the laboratory test values;
9. Participants with active hepatitis B or hepatitis C are allowed to be enrolled, provided that they receive strict antiviral therapy prior to medication and that liver function is adequate;
10. Syphilitic positive subjects are allowed to be enrolled, but strictly standardized anti-syphilis therapy is required before medication and syphilitic heart disease and other serious complications are excluded;
11. Fertile female subjects must have a negative serum pregnancy test at the time of screening and during at the end of the study; Male subjects whose partners are women of reproductive age should be surgically sterilized, or effective methods of contraception should be given during and at the end of the study;
12. Sign informed consent, voluntarily and be able to comply with the procedures of the trial and follow-up.

Exclusion Criteria:

1. Participating in a clinical study and receiving investigational drug therapy or investigational device within 4 weeks prior to initial dosing; If involved in non-interventional clinical trials can be included in this study;
2. There is unresectable or metastatic disease, pathology report showing microscopic positive surgical margin or extranodal invasion.
3. History of other malignancies within 5 years prior to the first dose of the study drug, except for malignancies that are expected to be cured after treatment (including but not limited to fully treated thyroid cancer, cervical carcinoma in situ, basal or squamous cell skin cancer, or ductal carcinoma in situ of the breast treated with radical surgery);
4. Previous treatment for NSCLC, including chemotherapy (preoperative chemotherapy treatment ≤ 2 cycles is allowed), targeted therapy (such as small molecule tyrosine kinase inhibitors targeting EGFR, ALK, VEGFR and other pathways, monoclonal antibodies, etc.), immunotherapy, investigational therapy, etc.;
5. The subject has undergone major surgery within 3 weeks prior to the first dose of the study drug (including primary tumor surgery, thoracotomy, laparotomy, excluding vascular access establishment procedures);
6. Use of traditional Chinese medicine and Chinese medicine preparations with anti-tumor treatment indications or auxiliary therapeutic effects on tumors within 14 days prior to the first dose of the study drug;
7. Received strong CYP3A inhibitors or inducers and narrow therapeutic index CYP3A substrates within 14 days before the first dose of the study drug;
8. Clinically significant cardiovascular diseases；
9. Severe active infection, interstitial lung disease / pneumonia, or any other serious underlying disease that may affect the subject's acceptance of protocol treatment within 2 weeks before the first dose;
10. Positive HIV antibody test result;
11. Active pulmonary tuberculosis;
12. Pregnant or lactating women;
13. Any other clinically significant disease or condition that the investigator believes may affect protocol compliance or the subject's signing of the informed consent form, or is not suitable for participating in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2029-01-15 (Estimated); Study Completion 2030-01-15 (Estimated)

PRIMARY OUTCOMES:
DFS | From enrollment to until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  From enrollment to until the date of first documented progression or date of death from any cause, whichever came first

SECONDARY OUTCOMES:
Adverse events | From enrollment to until the date up to 60 months
  adverse events using common terminology criteria for adverse events 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing cancer hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No